CLINICAL TRIAL: NCT06639841
Title: A Comparative Study on the Effectiveness of Virtual Reality-Facilitated Psychotherapy Vs. Yoga-Based Interventions for Managing Performance Anxiety Among Students
Brief Title: Effectiveness of Virtual Reality Psychotherapy and Yoga on Student Performance Anxiety
Acronym: VRvsHY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Collaborators: Romanian Academy (Other); Socola Institute of Psychiatry (Unknown)
Responsible Party: Principal Investigator, Marcel-Alexandru Gaina, Assistant Professor, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAR56-IRB-466/24; ICES 145/02.04.2024 (Registry Identifier: Scientific Council "Gheorghe Zane" Romanian Academy)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Performance Anxiety
Keywords: Performance anxiety; Students; Virtual Reality; Yoga; Psychotherapy
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model, where participants are divided into two distinct groups (arms). Each group will receive a different intervention simultaneously, without crossing over to the other group. The two arms will be independently assessed throughout the study period to compare the effects of the assigned interventions on the participants. This design allows for the direct evaluation of each intervention's impact, ensuring that comparisons can be made between the groups without overlap in treatment or intervention
Who Masked: Outcomes Assessor
Masking Description: Only the Outcomes Assessor will be blinded to the group assignments in this study. This masking is employed to avoid measurement bias when comparing the primary and secondary outcomes such that the assessor does not know whether the subject had a Virtual Reality (VR) intervention or Yoga. This approach improves the validity of data collection and measure outcomes.
  Because of the distinct and participatory nature of the interventions, VR and Yoga respectively, it is impossible to mask participants, care providers and researchers. This selective blinding approach of masking the Outcomes Assessor aims at an unbiased measure of outcome, despite the practical impossibility of full masking during behavioral and physical interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality facilitated Psychotherapy for Performance Anxiety (Experimental): Participants in this arm will undergo Virtual Reality (VR) facilitated Psychotherapy aimed to alleviate performance anxiety. The sessions will combine cognitive-behavioural therapy (CBT), exposure therapy and relaxation within VR environments. The program will be provided by a qualified integrative psychotherapist, 2-3 times per week, each lasting 30-60 minutes, over 4 weeks. The programme will be individualized for each participant, based on their anxiety levels and progression, including in-depth experiences to promote performance resilience.
  Interventions: Device: Virtual Reality Psychotherapy
- Yoga Training for Performance Anxiety (Experimental): Participants in this arm will undergo a Yoga-based intervention for performance anxiety. This therapy includes facilitated yoga sequences consisting of breathing (Pranayama), exercises (Asanas) and meditation, for body-mental relaxation. The course will be led by expert yoga instructors for 2x60 to 90 min sessions, twice per week, within 2 to 4 weeks. The trainers will focus on promoting mindfulness, reducing anxiety, and improving focus to help participants manage daily performance stressors.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Device: Virtual Reality Psychotherapy — Participants in this VR-facilited psychotherapy group will receive their treatment via Oculus Quest 2 and HTC Vive Flow wireless, standalone headsets systems to provide a comfortable immersive environment. The more hardware-intensive experiences will be carried out on Oculus Rift S headsets powered by high-end laptops.
  Sessions will last 30-60 minutes each, ranging from six to ten sessions within two to four weeks. The treatment will include reducing anxiety and improving emotion regulation through Cognitive-Behavioural techniques such as mindfulness, acceptance and commitement therapy, exposure therapy and 4-7-8 breathing. The same investigator will conduct all sessions to ensure uniformity. Additionally, subjects will undergo unsupervised VR at home with pre-programmed headsets to minimize investigator bias and maintain cosistancy of the relaxation and cognitive-behavioral strategies.
  Other Names: VRG
  Arms: Virtual Reality facilitated Psychotherapy for Performance Anxiety
Behavioral: Yoga — The Yoga group members will be guided in a yoga class focused on managing performance anxiety. The interventions will consist of body exercises (Asanas), breath (Pranayama) and meditation to increase relaxation, consciousness and resilience; typical yoga postures like Surya Namaskar, Padahastasana, Virabhadrasana, Bhujangasana and Shavasana will be included in the session, as will breathing movements like Ujjayi (Victory Breath).
  Each class will be 60-90 minutes long, and 6-10 classes will be taught in two to four weeks. The technique will be progressive, from the basic to more advanced postures as participants cultivate confidence and resilience. All classes will conclude with meditation to ease tension and cultivate mindfulness.
  Other Names: YG
  Arms: Yoga Training for Performance Anxiety

SUMMARY:
The goal of this pilot clinical trial is to compare two non-pharmacological interventions-Virtual Reality (VR) and Yoga techniques-in reducing performance anxiety in students aged 16-35. Performance anxiety, commonly experienced during public speaking and examinations, affects academic performance and well-being. The main questions it aims to answer are:

Does the VR-based guided meditation intervention reduce performance anxiety more effectively than Yoga-based relaxation techniques? Do participants experience better emotional regulation and improved quality of life with either intervention? Researchers will compare the VR intervention group to the Yoga intervention group to determine which intervention better alleviates anxiety symptoms and fosters improved emotional regulation during school performance.

Participants will:

Attend six to ten sessions of either VR-based guided meditation or Yoga-based relaxation over a period of four weeks.

Complete questionnaires to assess their anxiety levels, emotional regulation, and quality of life before and after the intervention.

DETAILED DESCRIPTION:
Detailed Description This randomized controlled trial (RCT) is designed to evaluate the comparative effectiveness of two non-pharmacological interventions-Virtual Reality (VR) and Yoga techniques-in reducing performance anxiety among students aged 16-35. Performance anxiety, a specific type of anxiety experienced in academic and public speaking situations, has a significant impact on students' academic performance and overall mental well-being. The study aims to explore accessible, non-invasive interventions that can be easily integrated into educational settings to help manage this condition.

The trial will compare VR-based guided relaxation and exposure therapy, delivered via the Guided Meditation VR software, with Yoga-based relaxation techniques, incorporating Hatha Yoga postures (asanas), breathing exercises (pranayama), and meditation (dhyana). Both interventions focus on providing mental relaxation, emotional regulation, and coping strategies to manage performance-related anxiety without the use of medications.

Rationale:

The choice of interventions is based on evidence supporting both VR and Yoga as effective tools for anxiety reduction. Virtual Reality has been shown to provide immersive environments that enhance relaxation, while allowing exposure to stressful situations in a controlled manner, which is crucial for performance anxiety. Guided Meditation VR enables students to practice mindfulness in virtual settings designed to reduce stress, using calming visuals and guided meditative exercises.

In contrast, Yoga is an ancient practice that has been widely studied for its ability to reduce anxiety through physical movement, controlled breathing, and meditation. By incorporating mindfulness and physical postures, Yoga may promote relaxation and help students improve their ability to regulate their physiological and emotional responses to anxiety-inducing situations.

Study Design:

The study will randomly assign participants to either a VR intervention group or a Yoga intervention group. Both interventions will be delivered over a period of 4 weeks, with 6-10 sessions, each lasting approximately 30-40 minutes. The interventions will be offered in a structured format, with the VR sessions focusing on mindfulness and relaxation in immersive environments, and the Yoga sessions integrating movement, breath control, and meditation.

Each participant's anxiety levels will be measured at baseline, immediately after the intervention, and during a follow-up period to assess the sustained effects of the interventions on anxiety reduction.

Virtual Reality Intervention:

The VR intervention will utilize the Guided Meditation VR software, accessible via VR headsets such as Oculus Quest 2 or HTC Vive Flow. The sessions will involve participants entering virtual environments specifically designed to promote relaxation and mindfulness, such as serene beaches, forests, and mountains. These environments are paired with guided meditation sessions aimed at calming the mind and reducing anxiety. Additionally, participants will be encouraged through guided imagery to engage in public speaking or exam scenarios, while using mindfulness techniques to reduce their anxiety responses. The immersive nature of VR allows participants to practice coping strategies in a safe, controlled setting.

Yoga Intervention:

The Yoga intervention will follow the principles of Hatha Yoga, focusing on practices that have been shown to promote relaxation and reduce anxiety. Sessions will incorporate a combination of physical postures (asanas), breath control exercises (pranayama), and meditation (dhyana). Participants will be guided through a series of gentle yoga postures aimed at reducing physical tension and promoting mental clarity. The breathing techniques and meditation components will focus on calming the mind and regulating the body's stress response, making this intervention particularly relevant for managing performance anxiety.

Feasibility and Acceptability:

In addition to the primary objective of reducing performance anxiety, this study will assess the feasibility and acceptability of integrating these interventions into student life. The ease of implementing VR and Yoga techniques in academic environments will be evaluated, as well as participant feedback on the usability and perceived effectiveness of each intervention.

Significance:

This trial addresses the growing need for accessible mental health interventions that can be seamlessly integrated into educational settings. By exploring the comparative benefits of Virtual Reality and Yoga, the study aims to provide insights into non-pharmacological treatments that may reduce the burden of anxiety on students. The results could inform future interventions that help students manage their mental health and academic performance more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years;
* Currently enrolled university students or recent graduates (within the last 2 years) pursuing further studies (e.g., Master's or PhD) in the same area of expertise;
* Mild to moderate levels of trait anxiety as measured by validated psychological inventories (e.g., STAI-Y1); Able to fully understand study procedures;
* No prior exposure to the specific interventions being tested (i.e., Virtual Reality Psychotherapy or Yoga interventions);
* Able to provide informed consent to participate in the study.

Exclusion Criteria:

* History of severe psychiatric disorders (e.g., schizophrenia, bipolar disorder);
* Currently receiving psychiatric or psychological treatment, including ongoing psychotropic medication;
* History of adverse reactions to Virtual Reality technology (e.g., motion sickness, dizziness, allergy to headset and controllers materials);
* Significant physical limitations preventing participation in yoga exercises;
* Pregnant individuals, due to physical limitations related to yoga and potential psychological sensitivity to Virtual Reality;
* Individuals not fluent in Romanian and English, as the interventions and assessments will be conducted in Romanian, with the Virtual Reality intervention partly in English.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-08 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Trait Anxiety Reduction | Measured 1 day before the first intervention session and within 1 day after the final intervention session of the program and also after major events such as faculty exams.
  The trait anxiety reduction will be measured with the Romanian validated version of the State-Trait Anxiety Inventory (STAI-Y2) Participant assessment: Previously trained and licensed STAI researchers will assess participants reported scores. The STAI-Y2 score ranges from 20 to 80, with higher scores indicating higher anxiety levels.

SECONDARY OUTCOMES:
State Anxiety Reduction | Measured at baseline, before each session, and 30 minutes after the interventions.
  We will assess state anxiety using the Romanian validated version of the State-Trait Anxiety Inventory (STAI-Y1); scores range from 20 to 80, with higher scores indicating higher levels of anxiety.
Emotional Regulation Strategies | Measured 1 day before the first intervention session and within 1 day after the final intervention session of the program.
  Emotional regulation strategies will be measured by the Emotion Regulation Questionnaire (ERQ), which measures two basic processes in emotional regulation: cognitive reappraisal and expressive suppression.
Quality of Life Improvement | Measured 1 day before the first intervention session and within 1 day after the final intervention session of the program.
  The quality of life will be measured through the Romanian population validated Quality of Life Inventory (QoLI) to reflect the participants' wellbeing and the impact of academic stress and anxiety. The scores will be assessed by a previously QoLi trained and licenced investigator.

OTHER OUTCOMES:
Performance Anxiety | Measured 1 day before the first intervention session and within 1 day after the final intervention session of the program.
  Measured using the Academic Anxiety Inventory for anxiety regarding particular academic assignments.
Qualitative Intervention Feedback | 60 minutes before and after each intervention.
  Through self-administered ratings of participants' comfort/discomfort with interventions at the end of each session, evaluations of effectiveness and overall perceptions of the Virtual Reality or Yoga intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel A Găină, Ass. Prof., Study Chair — University of Medicine and Pharmacy "Grigore T. Popa" Iași; Liviu A Măgurianu, Sci.Res.III, Study Director — Romanian Academy of Sciences "Gh. Zane" Institute Iasi
Locations (1):
- Romanian Academy of Sciences, Iași, Iaşi, Romania

IPD SHARING:
Plan to Share IPD: Yes
The IPD to be shared will consist of all anonymized information from the primary and secondary outcome measures, baseline information, and any other supporting data such as participant demographics. The data dictionaries, as well as any datasets supporting the published results will be distributed. These data will be available for future analysis, verification of the study results, or replication by other researchers.
  Time Frame:
  Access Criteria:
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting information will be published starting 6 months after the study results are published and will be available 2 years from the publication.
Access Criteria: Researchers who want to access the aforementioned data will need to make a formal request with a full scientific proposal outlining how the data will be used. The request will be reviewed by the external Data Safety and Monitoring Board (DSMB) review to verify that these requests are scientifically valid and ethical, in order to ensure participant data safety. The researchers who receive approval will have to sign a data-sharing contract regarding data protection within the specific utilization established terms.

REFERENCES:
- [Derived] Tofan CM, Magurianu LA, Axinte M, Gaina AM, Gaina M. Comparative Efficacy of Virtual Reality-Assisted Cognitive Behavioral Therapy Versus Yoga-Based Interventions for Reducing Performance Anxiety in Students: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 30;14:e66112. doi: 10.2196/66112. PMID 40587850